CLINICAL TRIAL: NCT06601764
Title: Effects Of Circuit Training and Progressive Resistance Exercise Program On Pulmonary And Physical Parameters In COPD Patients
Brief Title: Circuit and Resistance Training in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Zubair Khalid
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Circuit Training; Resistance Exercise; Pulmonary Function; Physical Function; Progressive Resistance Training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Circuit-Based Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Circuit training (Experimental): Circuits Training Exercise Group
  Interventions: Other: Circuit Training
- Group B: Progressive Resistance Exercise Group (Active Comparator): Progressive Resistance Exercise Group
  Interventions: Other: Progressive Resistance

INTERVENTIONS:
Other: Circuit Training — 1. Warm-up, balance
  2. Aerobic, balance
  3. Muscle strength Upper Limbs
  4. Muscle strength Lower Limbs
  5. Stretching both Upper Limb and Lower Limb
  Arms: Group A: Circuit training
Other: Progressive Resistance — 1. Muscle habituation exercises
  2. Hypertrophic phase 1 exercises
  3. Hypertrophic phase 2 exercises
  Arms: Group B: Progressive Resistance Exercise Group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is characterized by a combination of pulmonary and extra-pulmonary manifestations that directly contribute to the increase in exercise intolerance and dyspnea, especially in more advanced stages of the disease, leading to physical inactivity and consequent worsening of these signs and symptoms. COPD is a preventable and treatable lung disease. Solid evidence shows that physical training, the most important component of a Pulmonary Rehabilitation program (PR), reduces dyspnea and fatigue, increases exercise performance, and improves peripheral muscle strength, functional capacity, control of emotional function and quality of life of these patients' lives. Multicomponent physical training (MPT) proposes the performance of 3 or more components or physical training modalities within the same session and has demonstrated its benefits in several studies involving the elderly population. The main objective of the study will be to determine the effects of circuit training and resistive exercises on pulmonary function and physical parameters in population with COPD.

The study will be a randomized clinical trial and conducted for a duration of 09 months after the approval of synopsis. Data will be collected with Non-Probability Convenience Sampling Technique. A sample of 48 COPD patients will be recruited from DHQ Muzaffargarh. This will be a double blinded study with patients and assessor blinded to the intervention. COPD patients will be divided into two groups with group 1 treated with circuit training and group 2 treated with resistance exercise for duration of 10 weeks. Baseline values for Respiratory parameters and physical parameters will be collected and after 5 weeks and 10 weeks of treatment. Data will be analyzed using SPSS v 26. For within the group analysis Repeated Measure ANOVA will be used. For across the group analysis, independent sample T test will be used to compare the mean differences.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a progressive disease with deteriorating cardiopulmonary function that decreases the health-related quality of life (HRQL) and exercise capacity. Patients with COPD often have cardiovascular and muscular problems that hinder oxygen uptake by peripheral tissues, resulting in poor oxygen consumption efficiency. Only 20% of the estimated COPD cases are currently being identified and diagnosed in primary care in Pakistan.

Circuit training should be considered the most effective strategy to improve exercise capacity in patients with COPD. Supervision of the programs improves exercise capacity. Concerning strength outcome, the Circuit Training increased the strength of the upper and lower extremities. Only the magnitude of strength performance appears to be influenced by the training (number of sessions and frequency) and the training status. Moreover, low and moderate intensities and short rest time between exercises increase the magnitude of change in fat mass loss. Therefore, CT has been shown to be an effective method for improving body composition, cardio-respiratory fitness, and strength of the lower and upper limbs. Moreover, CT has been shown to elicit higher oxygen consumption during the session in comparison to a traditional strength-training session. Modalities of resistance training using elastic components presented similar effects on muscle strength, health status, exercise capacity, body composition and daily level of physical activity in individuals with COPD. The effects of elastic resistance were similar to conventional resistance training. CT significantly improves aerobic performance (i.e., increase maximum aerobic speed and aerobic performance) and VO2max (average 6.3%), showing that this type of training increases cardio-respiratory fitness independent of the training protocol. CT had an overall significant and large effect on upper (bench press) and lower strength (leg extension) performance (1-RM).only the magnitude of strength performance appears to be influenced by the training (i.e., number of sessions and frequency) and population characteristics (i.e., training status).

ELIGIBILITY:
Inclusion Criteria:

* Age range from 40 to 70 years
* Clinical -functional diagnosis of COPD criteria GOLD II and III
* Clinically stable (outside the period of exacerbation of the disease for at least 3 months),
* Independently able to perform instrumental activities of daily living, as assessed by the functional activities questionnaire
* No medical contraindications for physical exercise.

Exclusion Criteria:

* Pulmonary diseases such as asthma, pulmonary fibrosis, pneumonia and other non-pulmonary
* Sever or difficult to control ( heart disease or sequelae of acute or chronic orthopedic and/or neurological diseases),
* Those who use walking assist devices that could influence the exercise
* Enrolled in a physical training program within the last 3 months at baseline

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test | Baseline; 5th Week; 10th Week
  6MWT is a sub-maximal exercise test used to examine person aerobic capacity and endurance. This test initially developed to make an assessment of patient with cardiopulmonary issues. It is used to check the functional capacity of the individual and it provides useful information regarding all the body systems during physical activity, including cardiovascular and pulmonary system. It can used for all age group range 2 to above 64 years The test is easy to perfume , with standardized limited instructions and encouragement being given as person walk as far as possible over 6 minutes through a flat corridor. The final distance is recorded in meters.(
Pulmonary function test: Forced Vital Capacity (FVC) | Baseline; 5th Week; 10th Week
  The FVC is the forced vital capacity. It requires that the subject make a maximal inspiration to TLC, then make a maximal forced expiratory effort, leaving only the RV. In a normal subject, the FEV1/FVC is greater than 0.8; patients with obstructive lung disease, such as asthma or COPD, show a decreased FEV1/FVC
Pulmonary function test: Forced Expiratory Volume in 1 second (FEV1) | Baseline; 5th Week; 10th Week
  Forced expiratory volume (FEV1) calculates the amount of air that a person can force out of their lungs in 1 second. FEV1 values that are lower than average suggest the presence of COPD.
Pulmonary function test: FEV1/FVC Ratio | Baseline; 5th Week; 10th Week
  The FEV1/FVC ratio is a measurement of lung function that compares the forced expiratory volume in one second (FEV1) to the forced vital capacity (FVC). It's used to help diagnose and monitor lung conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Zubair Khalid, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabiliation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Priego-Jimenez S, Torres-Costoso A, Guzman-Pavon MJ, Lorenzo-Garcia P, Luceron-Lucas-Torres MI, Alvarez-Bueno C. Efficacy of Different Types of Physical Activity Interventions on Exercise Capacity in Patients with Chronic Obstructive Pulmonary Disease (COPD): A Network Meta-Analysis. Int J Environ Res Public Health. 2022 Nov 5;19(21):14539. doi: 10.3390/ijerph192114539. PMID 36361418
- [Background] Spielmanns M, Muller K, Schott N, Winkler A, Polanski H, Nell C, Boeselt T, Koczulla AR, Storre JH, Windisch W, Magnet FS, Baum K. [Impact of a Senso-Motoric Intervention in COPD-Patients Participating in an Outpatient Pulmonary Rehabilitation Program: A Randomized Controlled Trial]. Rehabilitation (Stuttg). 2017 Jun;56(3):159-166. doi: 10.1055/s-0042-119248. Epub 2017 Feb 23. German. PMID 28231596
- [Background] Mazzarin CM, Silveira BR, Lamezon AC, Cavon Luna B, Valderramas S. Effectiveness and Safety of Multicomponent Physical Training in Patients With Chronic Obstructive Pulmonary Disease: Protocol for a Randomized Clinical Trial. Health Serv Insights. 2023 May 2;16:11786329231169255. doi: 10.1177/11786329231169255. eCollection 2023. PMID 37153879
- [Background] Spielmanns M, Gloeckl R, Gropp JM, Nell C, Koczulla AR, Boeselt T, Storre JH, Windisch W. Whole-Body Vibration Training During a Low Frequency Outpatient Exercise Training Program in Chronic Obstructive Pulmonary Disease Patients: A Randomized, Controlled Trial. J Clin Med Res. 2017 May;9(5):396-402. doi: 10.14740/jocmr2763w. Epub 2017 Apr 1. PMID 28392859
- [Background] Chao KY, Liu WL, Nassef Y, Lai PZ, Wang JS. A pilot crossover trial assessing the exercise performance patients chronic obstructive pulmonary disease. Sci Rep. 2022 Mar 9;12(1):4158. doi: 10.1038/s41598-022-07698-z. PMID 35264615
- [Background] de Lima FF, Camillo CA, Grigoletto I, Uzeloto JS, Vanderlei FM, Ramos D, Ramos EMC. Effects of combining functional exercises with exercise training on daily physical activities and functionality in patients with COPD: a protocol for a randomized clinical trial. Trials. 2019 Dec 5;20(1):680. doi: 10.1186/s13063-019-3780-y. PMID 31805981
- [Background] Rinaldo N, Bacchi E, Coratella G, Vitali F, Milanese C, Rossi A, Schena F, Lanza M. Effects of Combined Aerobic-Strength Training vs Fitness Education Program in COPD Patients. Int J Sports Med. 2017 Nov;38(13):1001-1008. doi: 10.1055/s-0043-112339. Epub 2017 Oct 5. PMID 28982202